CLINICAL TRIAL: NCT04855669
Title: Effect of Embryo Migration After Embryo Transfer With Fresh Oocyte Donation Cycles on Pregnancy Outcomes
Brief Title: Effect of Embryo Migration in Fresh Oocyte Donation Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Turkan Gursu, Investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: YDU/2020/86-1239
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Infertility
Keywords: embryo migration; embryo transfer; fresh oocyte donation cycle; live birth rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to evaluate the impact of embryo distance from fundal endometrium, measured 60 minutes after transabdominal ultrasound guided embryo transfer(ET), on clinical pregnancy rates(CPR) and live birth rates(LBR) in fresh oocyte donation(OD) cycles.

DETAILED DESCRIPTION:
Embryos were considered to be staying at the initial expulsion site for long years. However, in 1976 Edwards and Steptoe reported a tubal ectopic pregnancy after in vitro fertilization (IVF) with a day-3 embryo transfer, which may be accepted as the earliest evidence for migration of embryos from the cavity. The migration concept is very recently taken into consideration by few authors, with studies on fresh IVF and frozen ET cycles.

Oocyte donation (OD) is a method of ART, in which by using young oocytes from donors the embryo quality is optimized. OD cycles have high LBRs, and are the choice of treatment in advanced reproductive age, repeated IVF failure, premature ovarian insufficiency(POI) and particular heritable genetic diseases. Donor oocytes can be used as fresh or cryoprotected-thawed, where fresh oocytes have higher LBRs.

In the literature, there are no studies performed in fresh OD cycles about air bubble and fundus distance after ET, and there are no studies performed whether there is any embryo migration after 60 minutes of ET and its effects on CPR and LBR.

Therefore, the investigators conducted this study to evaluate the impact of embryo distance from fundal endometrium, measured 60 minutes after transabdominal USG guided ET, on CPR and LBR in fresh OD cycles. In literature, this study is first to focus on embryo migration and LBR in fresh OD cycles.

ELIGIBILITY:
Inclusion Criteria:

* fresh oocyte donation cycles
* Anatomically anteverted-anteflexed recipient uterus
* partners with normal sperm parameters

Exclusion Criteria:

* Data of women who did not give approval
* IVF cycles
* frozen-thawed embryo transfer cycles
* cryopreserved-thawed OD cycles
* abnormal sperm parameters or need of any testicular interventions
* Anatomically retroverted-retroflexed recipient uterus
* teneculum required embryo transfers
* difficult transfers

Ages: 23 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — the study was performed with women who underwent embryo transfers
Study Population: The study included fresh OD cycles of recipient women.
Sampling Method: Non-Probability Sample
Enrollment: 653 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1 year
  In the literature, there are no studies performed in fresh OD cycles about air bubble and fundus distance after ET, and there are no studies performed whether there is any embryo migration after 60 minutes of ET and its effects on live birth rate outcome.

SECONDARY OUTCOMES:
clinical pregnancy rate | 1 year
  In the literature, there are no studies performed in fresh OD cycles about air bubble and fundus distance after ET, and there are no studies performed whether there is any embryo migration after 60 minutes of ET and its effects on clinical pregnancy and miscarriage rate outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Dunya In vitro fertilization center, Kyrenia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
After results are obtained we will decide.

REFERENCES:
- [Result] Saravelos SH, Wong AW, Chan CP, Kong GW, Cheung LP, Chung CH, Chung JP, Li TC. Assessment of the embryo flash position and migration with 3D ultrasound within 60 min of embryo transfer. Hum Reprod. 2016 Mar;31(3):591-6. doi: 10.1093/humrep/dev343. Epub 2016 Jan 11. PMID 26759141
- [Result] Ficicioglu C, Ozcan P, Kocer MG, Yesiladali M, Alagoz O, Ozkara G, Tayyar AT, Altunok C. Effect of air bubbles localization and migration after embryo transfer on assisted reproductive technology outcome. Fertil Steril. 2018 Feb;109(2):310-314.e1. doi: 10.1016/j.fertnstert.2017.10.032. Epub 2018 Jan 4. PMID 29306491
- [Result] Ozdemir AZ, Ayas B, Guven D, Turkmen A. Embryo flash migration in fresh and frozen embryo transfers for day 3 and day 5 embryos. Eur J Obstet Gynecol Reprod Biol. 2019 Jul;238:33-37. doi: 10.1016/j.ejogrb.2019.04.025. Epub 2019 May 4. PMID 31082741